CLINICAL TRIAL: NCT00371072
Title: Trabeculectomy With MMC Versus Ahmed Glaucoma Implant for Treatment of Pediatric Aphakic Glaucoma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8370
Record Dates: First submitted 2006-08-31; First posted 2006-09-01 (Estimated); Last update posted 2006-10-09 (Estimated); Status verified 2003-07

CONDITIONS: Pediatric Aphakic Glaucoma
Keywords: Aphakic Glaucoma; trabeculectomy with mitomycin- C; Ahmed glaucoma implant
MeSH Terms: interventions — Trabeculectomy; Mitomycin

INTERVENTIONS:
Procedure: trabeculectomy with mitomycin-C

SUMMARY:
In this randomized clinical trial we compare trabeculectomy with mitomycin-C (T+MMC) and Ahmed glaucoma implant (AGI) in treatment of aphakic glaucoma in children under 16 years of age.Complete and qualified success were defined as 5≤IOP≤21mmHg without and with medication respectively and we came to this point that; T+MMC and AGI are comparable in terms of success rate and complications in pediatric aphakic glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* congenital cataract
* history of cataract surgery
* under 16 years old
* Ocular pressure more than 21 mmHg

Exclusion Criteria:

* interruption of the follow up before 6 month
* Anterior segment dysgenesis

Ages: 0 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2004-03; Study Completion 2005-11

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Pakravan, MD, Principal Investigator — Ophthalmic Research Center of Shaheed Beheshti Medical University
Locations (1):
- Ophthalmic Research Center, Tehran, Tehran Province, Iran